CLINICAL TRIAL: NCT03294772
Title: Socio-health Impact of a Multifactorial Program of Hand Hygiene on Respiratory and Gastrointestinal Infections in Children Attending in Day-care Centres
Brief Title: Impact of a Multifactorial Program of Hand Hygiene on Infections in Children Attending in Day-care Centres
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación Biomédica Andalucía Oriental (Other)
Collaborators: Ministry of Health, Spain (Other Government)
Responsible Party: Principal Investigator, Ernestina Azor Martínez, Principal Investigador, Fundación Pública Andaluza para la Investigación Biomédica Andalucía Oriental
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FIBAO
Record Dates: First submitted 2017-09-15; First posted 2017-09-27 (Actual); Last update posted 2017-09-27 (Actual); Status verified 2017-09

CONDITIONS: Respiratory Tract Infections; Gastroenteritis
Keywords: Respiratory Tract Infections; gastroenteritis; hand sanitizer; handwashing; day care
MeSH Terms: conditions — Respiratory Tract Infections; Gastroenteritis | interventions — Hand Sanitizers; Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hand sanitizer group (Experimental): DCCs received alcohol-based hand sanitizer and a program educational. Characteristics of the hydroalcoholic gel (Alco aloe gel): chlorhexidine digluconate at 0.2% solution, phenoxyethanol 1%, benzalkonium chloride 0.1%. aloe barbadensis 5%, ethyl alcohol 70%, excipients c.s.p. 100 ml. Alcohol of between 70%, ph = 7-7,5.
  Interventions: Other: hand sanitizer
- Liquid soap group (Experimental): DCCs received soap and program educational. The liquid soaps used for handwashing in this study did not contain specific antibacterial component, ph= 5.5.
  Interventions: Other: liquid soap
- Control group (No Intervention): No hand sanitizer or educational program were used.

INTERVENTIONS:
Other: hand sanitizer — DCCs received alcohol-based hand sanitizer and a program educational.
  Other Names: educational intervention
  Arms: Hand sanitizer group
Other: liquid soap — DCCs received liquid soap and a program educational.
  Other Names: educational intervention
  Arms: Liquid soap group

SUMMARY:
It is well known that attending Day Care Centres (DCCs) can lead to an increase in the frequency of infections, due to the high incidence at this age and also the ease of transmission among children. This high incidence respiratory tract infections (RTIs) and acute gastroenteritis can also have a significant impact on the cost of health care systems, increasing the number of medical visits, hospitalizations and prescribing medications as symptomatic drugs or unnecessary antibiotics in some cases.The aim of the study was to determine whether a multifactorial hand-hygiene program (handwashing with soap and water vs hand sanitizer vs control group) reduce episodes due to RTIs and gastroenteritis in children attending DCCs. In addition, analyze the cost-effectiveness of these interventions.

DETAILED DESCRIPTION:
A randomized, controlled, and open study of 3 cohorts of families with children attending to DCCs, between the ages of 0 and 3, attending 25 DCC (911 children) in Almeria (Spain) was designed. This study was carried out over the course of 8 months (November 2013 to June 2014). A group of DCCs/families will perform hand hygiene with soap and water (SWG), another group with hand sanitizer gel (HSG) and a control group (CG) practiced usual handwashing techniques.

Intervention: The families and DCCs staff randomly assigned to HSG and SWG attended handwashing workshops of 2-hour duration. These took place one month before the beginning of the study. Workshop content included education about the most frequent infections in DCCs, their transmission, prevention, treatment, instructions on how and when hands should be washed, use of hand sanitizers and possible side effects in the HSG. Every 2 weeks, the research assistant and the teachers (staff) performed activities such as stories, songs and posters in the classroom, which are linked to hand hygiene and infection's transmission. In the Children/families in the HSG and SWG were instructed by the researchers, teachers, and research assistant to maintain the usual handwashing procedure after going to the toilet and when their hands were visibly dirty. They also were told to use the hand sanitizer and handwashing with water and liquid soap correctly in the following circumstances: after coming into the classroom; before and after lunch; after playing outside; when they went home; and after coughing; sneezing; or blowing their noses; after diapering.

Parents of the three groups completed the survey on sociodemographic characteristics and questions about hand hygiene referred to when and how their children wash their hands. Progenitors of children whit episodes due to RTIs and gastroenteritis collected the symptoms and handed in the completed form to the teacher. A research assistant collected the absence sheets of the participating classes weekly, called the parents of absent children to enquire about the cause of their absence, visited the classrooms and collaborated with the teachers in activities related to the hygiene of hands.

ELIGIBILITY:
Inclusion Criteria: Children between 0 and 3 years old enrolled in the aforementioned DCCs, attended the DCCs for at least 15 hours per week and whose parents/guardians had signed an informed consent document were included.

Exclusion Criteria: Children whit chronic illnesses or medication that could affect their likelihood of contracting an infection. Families who used hydroalcoholic gel prior to the start of the study and/or antiseptic soaps in the control group.

Ages: 4 Months to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 911 (Actual)
Dates: Start 2013-11-01 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2015-12-30 (Actual)

PRIMARY OUTCOMES:
the episodes due to respiratory tract infections | 8 moth
  The incidence rate of respiratory tract infections was calculated dividing the number of episodes due to tract respiratory infection by the number of pupils during the period of this study. Incidence rate ratio indicates (IRR): the ratio between incidence rate in 3 study groups
The episodes due to gastroenteritis | 8 month
  The incidence rate of gastroenteritis was calculated dividing the number of episodes due to gastroenteritis by the number of pupils during the period of this study. Incidence rate ratio indicates (IRR): the ratio between incidence rate in 3 study groups

SECONDARY OUTCOMES:
Antibiotic prescribing for respiratory infections | 8 month
  In this study presence or absence of at least 1 antibiotic prescription for each new episode of the RTIs (upper and low RTIs, otitis, amygdalitis, and bronchitis) was collected during the study period
The direct cost of respiratory and gastrointestinal infections | 8 month
  The direct costs of episodes due to respiratory and gastrointestinal infections were measured

IPD SHARING:
Plan to Share IPD: Yes
The researchers in this study have participated in: the study protocol, informed consent form, workshops on hand hygiene and transmission of infections and how to prevent it. They will also share statistical Analysis Plan and clinical study report
Supporting Information: SAP, CSR
Time Frame: Currently the database is available, we are waiting for statistical analysis

REFERENCES:
- [Derived] Azor-Martinez E, Garcia-Mochon L, Lopez-Lacort M, Strizzi JM, Munoz-Vico FJ, Jimenez-Lorente CP, Fernandez-Campos MA, Bueno-Rebollo C, Del Castillo-Aguas G, Balaguer-Martinez JV, Gimenez-Sanchez F. Child Care Center Hand Hygiene Programs' Cost-Effectiveness in Preventing Respiratory Infections. Pediatrics. 2021 Dec 1;148(6):e2021052496. doi: 10.1542/peds.2021-052496. PMID 34814193
- [Derived] Azor-Martinez E, Yui-Hifume R, Munoz-Vico FJ, Jimenez-Noguera E, Strizzi JM, Martinez-Martinez I, Garcia-Fernandez L, Seijas-Vazquez ML, Torres-Alegre P, Fernandez-Campos MA, Gimenez-Sanchez F. Effectiveness of a Hand Hygiene Program at Child Care Centers: A Cluster Randomized Trial. Pediatrics. 2018 Nov;142(5):e20181245. doi: 10.1542/peds.2018-1245. Epub 2018 Oct 8. PMID 30297500